CLINICAL TRIAL: NCT06227585
Title: Feasibility Study- REVEAL 475 System for Bevonescein-Assisted Intra-Operative Visualization of Nerves in Head and Neck Surgery
Brief Title: Feasibility Study for Bevonescein-Assisted Nerve Visualization in Head & Neck Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alume Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALM-488-003
Record Dates: First submitted 2023-11-16; First posted 2024-01-29 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Head and Neck Surgery
Keywords: parotidectomy; thyroidectomy; neck dissection; ALM-488; bevonescein; nerve; fluorescence; head and neck surgery; intra-operative; real-time; REVEAL 475

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Single Arm (Bevonescein) (Experimental): All patients will receive a single administration of bevonescein 500mg via IV infusion and the REVEAL 475 system will be used on all patients.
  Interventions: Device: REVEAL 475 System; Drug: Bevonescein

INTERVENTIONS:
Device: REVEAL 475 System — The REVEAL 475 system will be evaluated for its ability to visualize nerve-fluorescence following bevonescein administration.
Drug: Bevonescein — All patients will receive a single dose of bevonescein 500 mg via IV infusion 1-5 hours before surgery.
  Other Names: ALM-488

SUMMARY:
A feasibility study to evaluate the usability of the REVEAL 475 system in patients treated with bevonescein for nerve visualization during surgery.

DETAILED DESCRIPTION:
The REVEAL 475 system will be evaluated for its ability to visualize nerve-fluorescence following bevonescein administration. All patients will receive a single dose of bevonescein 500 mg via IV infusion 1-5 hours before undergoing parotidectomy, thyroidectomy or neck dissection surgery.

ELIGIBILITY:
Inclusion Criteria:

* Minimum of 16 years of age.
* Planning to undergo surgery in the Head and Neck.
* Study participant's primary surgical treatment is parotidectomy or thyroidectomy (unilateral or bilateral) or cervical neck dissection.
* Willing and able to provide written assent as required and written informed consent by a legally authorized representative after the nature of the study has been explained, and prior to any research-related procedures.
* Sexually active patients must be willing to use an acceptable method of contraception while participating in the study and for 30 days after receiving bevonescein.
* Females of childbearing potential must have a negative pregnancy test at screening and be willing to have additional pregnancy tests during the study.

Exclusion Criteria:

* Patient has a history of prior surgery and/or radiation to the intended surgical site.
* Patient has abnormal cardiac rhythm not controlled with medication.
* Patient has moderate to severe renal impairment as indicated by a glomerular filtration rate (GFR) < 60 mL/min.
* Patient has decreased hepatic function defined as AST/SGOT and ALT/SGPT that is higher than 20% of the institution's normal laboratory limits, and/or the patient has elevated total bilirubin that is higher than 20% of the institution's normal laboratory limits.
* Patient has unresolved acute toxicity from prior anti-cancer therapy, alopecia, neuropathy <= Grade 2, as well as other non-acute and stable anti-cancer therapy toxicities are acceptable.
* Patient has a history of fluorescein allergy.
* Patient has a history of drug-related anaphylactic or severe allergic reactions.
* Presense or history of any hypersensitivity to bevonescein or its excipients that, in the judgment of the Investigator, places the patient at increased risk for adverse effects.
* Presence of a concurrent disease or condition that may interfere with study participation including recent (within 6 months of screening) NYHA Class III or IV heart failure, myocardial infarction, or cerebrovascular accident.
* Presence or history of any condition, that in the view of the Investigator, places the patient at high risk of poor treatment compliance or of not completing the study.
* Pregnant or breastfeeding at screening or planning to become pregnant (self or partner) at any time during the study.
* Use of any investigational product or investigational medical device within 30 days prior to screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Surgeon perspective on REVEAL 475 system blue light illumination | Immediately after surgery
  Surgeon to provide responses to questions on a Likert scale 1-5 where a higher score means a better outcome
Surgeon perspective on REVEAL 475 system ease of use | Immediately after surgery
  Surgeon to provide responses to questions on a Likert scale 1-5 where a higher score means a better outcome

SECONDARY OUTCOMES:
Plasma concentration of bevonescein | 1.5-5 hours before surgery, during surgery, and 0-12 hours after surgery
  Measurement of the concentration of bevonescein in plasma from all patients immediately before, during and immediately after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Brett Berman, MD, Study Director — Chief Medical Officer
Locations (1):
- Jacobs Medical Center at UC San Diego Health, San Diego, California, United States